CLINICAL TRIAL: NCT03800407
Title: Pharmacokinetics of Anti-tuberculosis and Antiretroviral Drugs in Children
Brief Title: Contributing Factors for Poor HIV Treatment Response in Children With TB/HIV Coinfection
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201801820 TB/HIV - N; 2R01HD071779 (NIH); 5R01HD071779-10 (NIH)
Record Dates: First submitted 2019-01-03; First posted 2019-01-11 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Tuberculosis; Human Immunodeficiency Virus; Coinfection
Keywords: Pharmacokinetic; Concurrent antituberculosis therapy; Efavirenz; Virologic response; Children
MeSH Terms: conditions — Tuberculosis; Acquired Immunodeficiency Syndrome; Coinfection | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Ethylenediaminetetraacetic acid (EDTA) plasma and whole blood DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- EFV-based ART: ART-naïve HIV-infected children aged 3 - 14 years who initiate EFV-based ART
  Interventions: Other: Observational study
- Concurrent EFV-based ART plus anti-TB therapy: ART-naïve HIV-infected children aged 3 - 14 years with TB coinfection who initiate EFV-based ART while receiving first-line anti-TB therapy
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Outcome of EFV-based ART in children with TB/HIV coinfection compared to those with HIV only on EFV-based ART

SUMMARY:
Efavirenz (EFV)-based antiretroviral therapy (ART) remains the preferred regimen in human immunodeficiency virus (HIV)-infected children aged 3 years or older on rifampin-containing antituberculosis (anti-TB) therapy. This is because drug interactions between first-line anti-TB therapy with protease inhibitors (PIs) are more severe to adjust for, and interactions with integrase strand transfer inhibitors (INSTIs) are not well studied in that age group. Although, current weight-based EFV dosing recommendation is not optimal in some children, pharmacokinetic-treatment response (PK-PD) data to guide optimal dosing of EFV during concurrent rifampin-containing therapy in children is very limited. The study team propose that EFV concentrations outside the optimal therapeutic range in children will be associated with virologic failure due to lack of efficacy because of low concentrations or increased central nervous system (CNS) toxicities from high concentrations leading to poor medication adherence. The study will determine virological suppression rates in HIV-infected children with and without TB coinfection treated with standard efavirenz-based therapy and examine the factors contributing to poor virologic response.

DETAILED DESCRIPTION:
In a previous study, the study team found that first-line anti-TB therapy had minimal effect on EFV pharmacokinetics (PK) at the population level, but children with TB/HIV coinfection on anti-TB therapy had a trend towards worse virologic outcome compared to those with only HIV infection. Due to the small sample size, the study team were unable to examined the patient factors contributing to the poor virologic response. The study team hypothesized that virologic suppression rates on EFV-based therapy is significantly lower in children with TB/HIV coinfection compared to those with HIV alone. In addition, virologic response will be dependent EFV plasma concentrations, CYP2B6 516 G>T genotype and/or adherence level. This hypothesis is based on the premise that extremes (low and high EFV concentration, respectively) could lead to virologic failure because of lack of efficacy or intolerable side effects leading to poor adherence. The current study will investigate the effect of anti-TB therapy, CYP2B6 genotype and pharmacokinetically determined adherence level on virologic response in children with TB/HIV coinfection treated with EFV-based ART.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive children with or without active TB
* Antiretroviral-naïve to efavirenz and meet criteria for initiation or switch to efavirenz-based ART
* Are available for follow-up until achievement of a study endpoint like completion of study at 6 months or discontinuation of ART.

Exclusion Criteria:

* Unable to obtain informed signed consent parent(s) or legal guardian
* Have AIDS-related opportunistic infections other than TB
* History of acute hepatitis within 30 days of study entry
* Persistent vomiting or diarrhea at time of enrolment
* Hemoglobin < 6 g/dl, white blood cells < 2500/mm3, serum creatinine > 1.5 mg/dl, aspartate transaminase (AST) and alanine transaminase (ALT) > 2 times upper limit of normal

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 3 to 14 years old with HIV infection with or without active TB
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
TB coinfection status and HIV RNA < 200 copies/mL on EFV-based ART in HIV-infected children. | At week 24 of HIV therapy.
  The proportion of children with TB/HIV coinfection with virological suppression (HIV RNA < 200 copies/mL) on EFV-based ART and anti-TB therapy compared to that in children with only HIV infection on EFV-based therapy.

SECONDARY OUTCOMES:
Efavirenz plasma mid-dose concentration and HIV RNA suppression < 200 copies/mL. | Up to week 24 of HIV therapy.
  Relationship between EFV mid-dose concentration and HIV RNA suppression rate in the combined population of HIV-infected children with and without TB coinfection.
Random efavirenz concentration below the limit of detection (poor ART adherence) and HIV RNA suppression rate. | Up to week 24 of HIV therapy.
  Relationship poor ART adherence and EFV-based ART response in the combined population of HIV-infected children with and without TB coinfection.
CYP2B6 516G>T genotype status and random efavirenz concentration below the limit of detection (poor ART adherence). | Up to week 24 of HIV therapy.
  Relationship between CYP2B6 516G>T genotype status and likelihood of poor EFV-based ART adherence.
CYP2B6 516G>T genotype status and HIV RNA suppression < 200 copies/mL. | Up to week 24 of HIV therapy.
  Relationship between CYP2B6 516G>T genotype status and likelihood of HIV RNA suppression.
TB coinfection status and risk of virological failure on EFV-based ART. | Up to week 48 of HIV therapy.
  Proportion of children with TB/HIV coinfection compared to those with only HIV infection with virological failure (HIV RNA > 1000 copies/mL) at 12 months of EFV-based ART.

CONTACTS AND LOCATIONS:
Overall Officials: Awewura Kwara, MD, Principal Investigator — University of Florida
Locations (1):
- Kwame Nkrumah University of Science and Technology, Kumasi, Ghana

IPD SHARING:
Plan to Share IPD: Undecided